CLINICAL TRIAL: NCT03566706
Title: Parents' View About Discussing Health Behaviors With Their Children
Brief Title: Parents' View About Discussing Health Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Responsible Party: Principal Investigator, Linda Diane Cameron, Professor, University of California, Merced
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: UCM2018-36
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Parents of Children Ages 10 to 17 Years Old

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unhealthy Eating (Experimental)
  Interventions: Behavioral: Discussion Tool: Unhealthy Eating
- Marijuana Use (Experimental)
  Interventions: Behavioral: Discussion Tool: Marijuana Use
- Sedentary Behavior (Experimental)
  Interventions: Behavioral: Discussion Tool: Sedentary Behavior

INTERVENTIONS:
Behavioral: Discussion Tool: Unhealthy Eating — Parents will randomly be assigned to one of three discussion tools that will provide parents with tools on how to communicate with their children about unhealthy eating, marijuana use, or sedentary behavior.
  Other Names: Parent Discussion Tools
  Arms: Unhealthy Eating
Behavioral: Discussion Tool: Marijuana Use — Parent Discussion Tools
  Arms: Marijuana Use
Behavioral: Discussion Tool: Sedentary Behavior — Parent Discussion Tools
  Arms: Sedentary Behavior

SUMMARY:
It is important to increase understanding of parent views about discussions of health risk behaviors with their children, in order to guide efforts to develop health communication strategies aimed at promoting parent and child discussion of these behaviors. In turn, this may lead to a decrease in youth engaging in health-risk behaviors. This study explores parental views about discussing health risk behaviors with their children and then tests the effects of a discussion tool on parents conversations with their children about unhealthy eating, marijuana use, and sedentary behavior. Participants will include parents living in the United States who have children ages 10 to 17 years old.

DETAILED DESCRIPTION:
Adolescence is often characterized as a particularly difficult time for children. Though adolescents begin to desire independence from their parents, parents still play an integral role in prevention of health-risk behaviors in their children. In fact, the quality of the parent-child relationship continues to serve as a determining factor of whether or not an adolescent will engage in harmful behaviors. Often times, this may lead to the practice of risky and harmful behaviors, such as, poor diet, substance use, unprotected sex, and reckless driving. The quality of the parent-child relationship continues to serve as a determining factor of whether or not an adolescent will engage in harmful behaviors. For instance, weekly parent-child discussions have also been identified as one of the strongest factors in influencing healthier food choices in adolescents. It is important to increase understanding of parent views about discussions of health risk behaviors with their children, in order to guide efforts to develop health communication strategies aimed at promoting parent and child discussion of these behaviors. In turn, this may lead to a decrease in youth engaging in health-risk behaviors.

This study explores parental views about discussing health risk behaviors with their children and then tests the effects of a discussion tool on parents conversations with their children about unhealthy eating, marijuana use, and sedentary behavior. Participants will include parents living in the United States who have children ages 10 to 17 years old. The study will consist of a baseline survey, and then a follow-up survey four weeks later. Participants will be randomly assigned to one of three discussion tool conditions that include marijuana use, unhealthy eating, or sedentary behavior. One month later, participants will be invited to complete a follow-up survey that will measure discussion behavior, followed by items from the initial survey. Following the survey completion, participants will read a brief explanation of the study and receive links to websites of national health organizations with information about unhealthy eating and marijuana use.

ELIGIBILITY:
Inclusion Criteria:

* Parent of children ages 10 to 17 years old living in the United States.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Intentions | 4 weeks
  The measure of parental intentions to discuss unhealthy eating and marijuana use with their child, adapted from established measures of behavioral intentions (Ajzen, 2002; Gibbons & Gerrard, 1995), included six items, 3 for unhealthy eating, and 3 for marijuana use. The measure began with the stem: "In the next four weeks, to what extent do you plan to discuss unhealthy eating (or marijuana use) with your child?," "In the next four weeks, to what extent will you try to discuss unhealthy eating (or marijuana use) with your child?," and "In the next four weeks, how likely is it that you will discuss unhealthy eating (or marijuana use) with your child?" Ratings ranged from 1 (not at all) to 5 (definitely).
Willingness | 4 weeks
  This measure was adapted from measures used to assess similar constructs such as within the context of cigarette smoking (Gibbons & Gerrard, 1995). The measure of parental willingness to discuss unhealthy eating and marijuana use with their child included the following stems: "Your child wants to attend a party in four weeks where there would be unhealthy foods (such as, soda, fried foods, chips, candy, ice cream, etc.) (or marijuana). How willing would you be to ask your child to not attend the party within the next four weeks?" "How willing would you be to discuss unhealthy eating (or marijuana use) with your child over the next four weeks?" and "How willing would you be to discuss potential concerns about unhealthy eating (or marijuana use) with your child over the next four weeks?" Ratings ranged from 1 (very unwilling) to 5 (very willing).
Discussion | 4 weeks
  Participant discussion behavior will be measured in the follow-up survey with 4 items, "Since the last session four weeks ago, did you talk about unhealthy eating (or marijuana use or sedentary behavior) with your child?" Participant will respond with a no (0) or yes (1). If participant answered yes, they will be able to briefly describe what they said to their child for all three conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Merced, Merced, California, United States